CLINICAL TRIAL: NCT02319447
Title: Increasing Kidney Transplant Among Blacks on the Transplant Waiting List
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Barnabas Medical Center (Other)
Collaborators: University of California, Los Angeles (Other); Rutgers University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SBMC 2012-69; R01DK098744 (NIH)
Record Dates: First submitted 2014-12-15; First posted 2014-12-18 (Estimated); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Chronic Kidney Disease; End-Stage Renal Disease
Keywords: Living Donation; Kidney Transplantation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): After randomization, these study participants will receive the Usual Care received by all listed kidney transplant candidates at our center.
- Additional education (Experimental): These study participants will be invited to attend a 60-90 minute educational seminar, entitled Destination: Transplant, delivered in a group setting. They will also receive monthly mailings for 9 months and a follow-up phone call from a transplant educator.
  Interventions: Behavioral: Additional education

INTERVENTIONS:
Behavioral: Additional education — Our Intervention includes a 60-90 minute educational seminar, entitled "Destination: Transplant", featuring "live" speakers, delivered to small groups of Black kidney transplant candidates and their family and friends. Topics include: 1) basic facts about Chronic Kidney Disease (CKD), transplant, and the waiting list; 2) the experience of receiving a LDKT transplant (by a Black LDKT recipient); 3) the experience of serving as a living kidney donor (by a Black living kidney donor); and 4) strategies to increase the chances of getting a transplant sooner. Participants receive monthly mailed, written information for 9 months and a follow-up phone call from a transplant educator, 3 months after attending the seminar.
  Arms: Additional education

SUMMARY:
For most patients with kidney failure, living donor kidney transplant (LDKT) is their best treatment option. Unfortunately, Blacks (vs. non-Blacks) are more likely to have kidney failure but less likely to receive LDKTs. In this study, the investigators will test an intervention designed to address this disparity, by performing a parallel group, two-arm randomized clinical trial among 500 Black kidney transplant candidates. The main objective of this study is to test an educational and behavioral intervention that is designed to increase receipt of LDKT among transplant candidates (persons active on the deceased donor kidney transplant waiting list) who are Black. Our overall hypothesis is that a multi-component intervention administered to Black transplant candidates will increase both readiness to pursue LDKT and actual receipt of LDKTs. The investigators will randomly assign kidney transplant candidates on the kidney transplant waiting list to either: (1) a control group that will receive Usual Care, or (2) an Intervention group that will receive a group-based intervention, as well as monthly mailings and a follow-up phone call by a transplant educator.

DETAILED DESCRIPTION:
The best treatment for severe chronic kidney disease is usually a living donor kidney transplant (LDKT), but large racial disparities persist in receipt of LDKTs. In 2011, Blacks, who comprised 36.8% of the dialysis population, received 32.2% of deceased donor kidney transplants (DDKTs) but just 14.0% of LDKTs. Among kidney transplant candidates who are Black, their lower rate of LDKT largely stems from a lack of donor volunteers (persons interested in donating a living kidney to them). The most effective ways to motivate and help Black transplant candidates to "recruit" or identify any (or more) donor volunteers remain unclear. Several interventions appear promising and are being tested, but none has proven both practical and effective.

Transplant candidates, particularly those who are Black, report that multiple barriers prevent them from receiving LDKTs. These barriers include minimal knowledge about LDKT; fears about donors' future health; guilt; medical mistrust; and discomfort about how to discuss LDKT with family and friends. Most transplant candidates have never met either a kidney donor or a recipient of a transplant or LDKT. A multi-component intervention that efficiently addresses these barriers could plausibly increase receipt of LDKT among Blacks.

The main objective of this study is to test an educational and behavioral intervention that is designed to increase receipt of LDKT among transplant candidates (persons active on the DDKT waiting list) who are Black. Our overall hypothesis is that a multi-component intervention administered to Black transplant candidates will increase both readiness to pursue LDKT and actual receipt of LDKTs.

To meet this objective and test our hypothesis, we propose a two-arm, parallel group randomized trial among 500 Black kidney transplant candidates. After Black transplant candidates are placed on the waiting list for a DDKT, we will randomize them to either: (1) a control group that will receive Usual Care, or (2) an Intervention group that will receive a group-based intervention as well as monthly mailings and a follow-up phone call by a transplant educator. Participants randomized to the Intervention will be asked to attend, in small groups with any family and friends, a 60-90 minute seminar that will feature brief talks regarding: ●basic facts about CKD, transplant, and the waiting list; ●the experience of receiving a LDKT transplant (by a Black LDKT recipient); ●the experience of serving as a living kidney donor (by a Black living kidney donor); and ●strategies to increase the chances of getting a transplant sooner.

Our Specific Aims are as follows:

Aim 1 (Primary Aim): To compare readiness to pursue LDKT and receipt of LDKT in the Intervention vs. Usual Care groups of our randomized clinical trial, during the 18 months after randomization

Hypothesis: Exposure to the multi-component Intervention is associated with an increase in readiness to pursue LDKT and an increase in receipt of LDKT

Aim 2: To determine the baseline social and behavioral variables that modify the effect of the Intervention upon readiness to pursue LDKT and actual receipt of LDKT

Hypothesis: Greater knowledge of LDKT and greater readiness to pursue LDKT are associated with receipt of LDKT

Aim 3: To determine whether changes in social and behavioral variables mediate the effects of the Intervention upon readiness to pursue LDKT and actual receipt of LDKT

Hypothesis: Increases in readiness to pursue LDKT are associated with receipt of LDKT

ELIGIBILITY:
Inclusion Criteria:

* self-reported as Black or African-American
* 21 years of age or older
* active on kidney transplant waiting list at Saint Barnabas Medical Center

Exclusion Criteria:

* limited English proficiency
* unable or unwilling to provide informed consent
* unable to complete in-person and telephone questionnaires (including hearing impairment or low vision)
* lack a working telephone
* live 150 miles or greater from transplant center
* enrolled in prior randomized intervention trial, NCT01261910, at our center
* currently already scheduled to receive a live donor kidney transplant
* active on the simultaneous pancreas-kidney transplant waiting list

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2014-12; Primary Completion 2018-02 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change in readiness to pursue LDKT at 9 months | Baseline, 9 months
  Our primary outcome is the proportion of study participants with an increase in their readiness to pursue LDKT. Readiness to pursue LDKT is assessed by the patient's Stage of Change regarding pursuing live donation, based upon James Prochaska's Transtheoretical Model. The Stages of Change regarding pursuit of living donation include: not considering (Pre-contemplation), considering (Contemplation), preparing to pursue (Preparation), or taking action to pursue (Action) living donation within the next 6 months. Stage of Change will be assessed at baseline and at 9 months post-baseline.

SECONDARY OUTCOMES:
Receipt of a LDKT | 18 months
  Among trial participants, we will determine whether or not they received a LDKT in the United States during the 18 months after they were enrolled in the trial and randomized. This determination will be made by examining each study participant's medical records.
Number of donor volunteers recruited and evaluated | 18 months
  We will examine each study participant's medical records to determine how many living donor volunteers contacted the transplant center to donate and how many donor volunteers were evaluated by the transplant center, during the 18 month follow-up period.
Status on kidney transplant waiting list | 18 months
  After 18 months of follow-up, for study participants who remain on the waiting list, we will determine whether they are: ●active (Status 1), or ●inactive (Status 7) on the waiting list. Other patients will have been removed from the Saint Barnabas Medical Center (SBMC) waiting list because they: ●died; ●became too sick to transplant; ●refused transplant; ●transferred to another center; ●improved and no longer required transplant; ●received a DDKT; ●received a LDKT; or ●other. We will determine these reasons, along with the date they occurred, by examining the medical records for each patient.
Change in knowledge of LDKT at 9 months | Baseline, 9 months
  We will assess knowledge of transplant and LDKT at baseline and 9 months, using a questionnaire containing multiple-choice and true-false questions.

OTHER OUTCOMES:
Change in knowledge of LDKT at 1 week post-intervention | Baseline, 1 week post-intervention
  We will assess knowledge of transplant and LDKT using a questionnaire containing multiple-choice and true-false questions. Each patient in the Usual Care arm will be matched to a patient in the Intervention arm. One week after attending the Intervention, each patient in the Intervention arm and the Intervention patient's matched Usual Care patient will have their knowledge of LDKT assessed. We will compare this score to the score obtained at baseline.
Change in readiness to pursue LDKT at 1 week post-intervention | Baseline, 1 week post-intervention
  We will measure an increase in study participants' readiness to pursue LDKT, assessed by their Stage of Change regarding pursuing living donation, based upon James Prochaska's Transtheoretical Model. The Stages of Change regarding pursuit of live donation include: not considering (Pre-contemplation), considering (Contemplation), preparing to pursue (Preparation), or taking action to pursue (Action) living donation within the next 6 months. Each patient in the Usual Care arm will be matched to a patient in the Intervention arm. One week after attending the Intervention, each patient in the Intervention arm and the Intervention patient's matched Usual Care patient will have their Stage of Change assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Francis L Weng, MD, MSCE, Principal Investigator — St. Barnabas Medical Center
Locations (1):
- Saint Barnabas Medical Center, Livingston, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-22): https://cdn.clinicaltrials.gov/large-docs/47/NCT02319447/Prot_SAP_000.pdf